CLINICAL TRIAL: NCT04065295
Title: A Randomised, Single-blind, Placebo-controlled Trial in Parallel Group Design to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses of BI 1356225 Administered as Oral Solution and Tablets to Healthy Male Subjects, and a Randomised, Open-label, Single-dose, Two-way Cross-over Bioavailability Comparison of BI 1356225 as Tablet With and Without Food
Brief Title: A Study to Test How Well Healthy Men Tolerate Different Doses of BI 1356225
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1427-0001; 2019-000198-22 (EudraCT Number)
Record Dates: First submitted 2019-08-21; First posted 2019-08-22 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Rising Dose Part (Experimental)
  Interventions: Drug: BI 1356225; Drug: Placebo
- Bioavailability Part (Experimental)
  Interventions: Drug: BI 1356225

INTERVENTIONS:
Drug: BI 1356225 — Oral Dose
Drug: Placebo — Oral dose
  Arms: Single Rising Dose Part

SUMMARY:
The main objectives of the SRD part of this trial are to investigate safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of BI 1356225 in healthy male subjects following oral administration of single rising doses. The main objective of the BA part of this trial will be to explore the influence of food on the bioavailability of tablet fasted versus tablet fed

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
* Age of 18 to 45 years (inclusive)
* BMI of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with GCP and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* Further exclusion criteria apply

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
The primary endpoint for assessment of safety and tolerability of BI 1356225 is the percentage of subjects with drug-related adverse events (both trial parts) | Up to 30 days

SECONDARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | Up to 30 days
Cmax (maximum measured concentration of the analyte in plasma) | Up to 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: http://trials.boehringer-ingelheim.com/